CLINICAL TRIAL: NCT03788408
Title: Effects of Intensive Psychotherapy and Case Management for Karen Refugees in Primary Care: A Randomized Control Trial
Brief Title: Intensive Psychotherapy and Case Management for Karen Refugees in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Center for Victims of Torture, United States (Other)
Collaborators: University of Minnesota (Other); HealthEast Care System (Other)
Responsible Party: Principal Investigator, Maria Vukovich, Research Associate, The Center for Victims of Torture, United States
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2018-12-20; First posted 2018-12-27 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Delivery of Intensive Behavioral Services to Refugees in Primary Care
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Psychotherapy Case Management (Experimental): Treatment group received Intensive Psychotherapy and Case Management (IPCM) delivered by psychotherapists and social worker with expertise in refugee trauma and mental health.
  Interventions: Behavioral: Intensive Psychotherapy and case management for refugee trauma
- Treatment as Usual (TAU) (Active Comparator): Treatment as Usual group received ongoing care from their primary care providers without the involvement of CVT (except for the collection of outcomes). TAU patients could be referred to a full range of outpatient and community-based behavioral health services by their primary care physician.
  Interventions: Behavioral: Intensive Psychotherapy and case management for refugee trauma

INTERVENTIONS:
Behavioral: Intensive Psychotherapy and case management for refugee trauma — CVT's approach emphasized active interdisciplinary coordination and a relational focus anchored in cultural humilityX to address survivors' priorities, empower survivors as the primary architects of their healing, and work alongside each survivor to co-construct meaning and behavioral change.

SUMMARY:
Patients in the IPCM group (n = 112) received intensive psychotherapy and case management, and those in the CAU group (n = 102) received care as usual, including behavioral health referrals and/or brief onsite interventions.

DETAILED DESCRIPTION:
IPCM patients received routine services from both a psychotherapist and separate mental health case manager for one year; duration of each appointment was 45 minutes - 1 hour; frequency of appointments was weekly or every other week, dependent on participant availability. A face-to-face professional interpreter was utilized unless the CVT provider was a native Karen speaker.

Participants in the control group received care as usual, without CVT involvement other than administration of the outcome measures. Once randomized, CAU patients could be referred to a full range of outpatient and community-based behavioral health services by their primary care physician.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria included Major Depression diagnosis by SCID interview, Karen refugee, ages 18-65.

Exclusion Criteria:

* Exclusion criteria were current participation in individual psychotherapy or case management, psychosis, or substance use problems on the CAGE-AID.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Depression over time | Collected at baseline, 3, 6, and 12 months
  Hopkins Symptom Trauma Checklist (HSCL-25) consists of 25 items with 15 items evaluating depression symptoms with response scale scores ranging from 1 (not at all) to 4 (extremely) indicating the frequency and severity of symptoms. Low scores indicate low symptoms while higher scores indicate greater symptoms of depression.
Change in Anxiety over time | Collected at baseline, 3, 6, and 12 months
  Hopkins Symptom Trauma Checklist (HSCL-25) consists of 25 items with 10 items assessing anxiety symptoms with response scale scores ranging from 1 (not at all) to 4 (extremely) indicating the frequency and severity of symptoms. Low scores indicate low symptoms while higher scores indicate greater symptoms of anxiety.
Change in PTSD over time | Collected at baseline, 3, 6, and 12 months
  Posttraumatic Stress Disorder (PDS-5) consists of 21 items evaluating symptoms of posttraumatic stress with response scale scores ranging from 1 (not at all) to 4 (extremely) indicating the frequency and severity of symptoms. Low scores indicate low symptoms while higher scores indicate greater symptoms of PTSD.
Change in Pain over time | Collected at baseline, 3, 6, and 12 months
  Pain Complaints Scale consists of 5 items assessing general pain symptoms with response scale scores ranging from 1 (not at all) to 4 (extremely) indicating the frequency and severity of symptoms. Low scores indicate low symptoms while higher scores indicate greater symptoms of pain.
Change in Safety/Basic Needs over time | Collected at baseline, 3, 6, and 12 months
  Social Circumstances and Social Functioning Inventory (SCFI-37), consists of 37 items that measure adaptive social functioning in 6 subscales (safety/basic needs, immigration stability, employment, social support, cultural adjustment and community engagement) with response scale scores ranging from 0 (low functioning) to 4 (high functioning). Safety/basic needs measures frequency and quality of basic needs met in housing, clothing, food, and transportation. Subscale scores are calculated as total scores.
Change in Immigration Stability over time | Collected at baseline, 3, 6, and 12 months
  Social Circumstances and Social Functioning Inventory (SCFI-37), consists of 37 items that measure adaptive social functioning in 6 subscales (safety/basic needs, immigration stability, employment, social support, cultural adjustment and community engagement) with response scale scores ranging from 0 (low functioning) to 4 (high functioning). Immigration stability measures legal status and stability for work, healthcare and residence in the country and progress towards citizenship. Subscale scores are calculated as total scores.
Change in Employment over time | Collected at baseline, 3, 6, and 12 months
  Social Circumstances and Social Functioning Inventory (SCFI-37), consists of 37 items that measure adaptive social functioning in 6 subscales (safety/basic needs, immigration stability, employment, social support, cultural adjustment and community engagement) with response scale scores ranging from 0 (low functioning) to 4 (high functioning). Employment subscale consists of 5 items measuring motivation for, and frequency and quality of employment. Subscale scores are calculated as total scores.
Change in Social Support over time | Collected at baseline, 3, 6, and 12 months
  Social Circumstances and Social Functioning Inventory (SCFI-37), consists of 37 items that measure adaptive social functioning in 6 subscales (safety/basic needs, immigration stability, employment, social support, cultural adjustment and community engagement) with response scale scores ranging from 0 (low functioning) to 4 (high functioning). The social support subscale consists of 5 items measuring frequency and quality of social connections in family and friends. Subscale scores are calculated as total scores.
Change in Cultural Adjustment over time | Collected at baseline, 3, 6, and 12 months
  Social Circumstances and Social Functioning Inventory (SCFI-37), consists of 37 items that measure adaptive social functioning in 6 subscales (safety/basic needs, immigration stability, employment, social support, cultural adjustment and community engagement) with response scale scores ranging from 0 (lower functioning) to 4 (higher functioning). Cultural Adjustment consists of 5 items measuring adaptation to new cultural and geographic community.
  Subscale scores are calculated as total scores.
Change in Community Engagement over time | Collected at baseline, 3, 6, and 12 months
  Social Circumstances and Social Functioning Inventory (SCFI-37), consists of 37 items that measure adaptive social functioning in 6 subscales (safety/basic needs, immigration stability, employment, social support, cultural adjustment and community engagement) with response scale scores ranging from 0 (low functioning) to 4 (high functioning). Community engagement consists of 6 items measuring participation in civic, political, social and educational activities in the geographic community. Subscale scores are calculated as total scores.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vukovich M, Esala J, Beckman A, Northwood A, Vinson G, Letts J, Danner C. Cost Savings from Integrating Behavioral Health in Primary Care: A Pragmatic Randomized Control Trial with Karen Refugees. J Immigr Minor Health. 2025 Nov 2. doi: 10.1007/s10903-025-01806-7. Online ahead of print. PMID 41176745
- [Derived] Northwood AK, Vukovich MM, Beckman A, Walter JP, Josiah N, Hudak L, O'Donnell Burrows K, Letts JP, Danner CC. Intensive psychotherapy and case management for Karen refugees with major depression in primary care: a pragmatic randomized control trial. BMC Fam Pract. 2020 Jan 28;21(1):17. doi: 10.1186/s12875-020-1090-9. PMID 31992234